CLINICAL TRIAL: NCT04655911
Title: A Long-term Follow-up Study of Patients With MPS IIIB From Gene Therapy Clinical Trials Involving the Administration of ABO-101 (rAAV9.CMV.hNAGLU)
Brief Title: A Long-term Follow-up Study of Patients With MPS IIIB Treated With ABO-101
Status: Terminated | Type: Observational
Why Stopped: Abeona has decided to discontinue development activities for Product AB0-101 due to a lack of drug supply and for business reasons unrelated to the product safety profile and/or signs of efficacy
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LTFU-ABO-101; 2019-002936-97 (EudraCT Number)
Record Dates: First submitted 2020-11-17; First posted 2020-12-07 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Mucopolysaccharidosis III-B
Keywords: MPS IIIB; Mucopolysaccharidosis IIIB; Sanfilippo B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ABO-101: Participants from prior interventional trials involving the administration of ABO-101.
  Interventions: Biological: ABO-101

INTERVENTIONS:
Biological: ABO-101 — Gene therapy rAAV9.CMV.hNAGLU

SUMMARY:
This is a multicenter, non-interventional, long-term follow-up (LTFU) study in participants who have been treated with ABO-101 in a prior trial. Eligible participants will undergo clinical evaluations at prespecified intervals for 3 years from the last visit in the prior clinical trial (up to 5 years post-treatment).

DETAILED DESCRIPTION:
This is a multicenter, noninterventional, long-term follow-up study of patients with (Mucopolysaccharidosis IIIB) MPS IIIB who have completed a prior clinical trial involving the administration of ABO-101. This study is designed to provide LTFU in accordance with the FDA and European Medicines Agency (EMA) guidelines for patients treated with gene therapy products. The duration of the current study is 3 years for a total of up to 5 years post-treatment for these participants who rollover from a prior clinical trial of ABO-101. Participants will have a maximum of 5 annual scheduled visits with assessments as specified in the schedule of assessments.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have completed a prior clinical trial involving the administration of ABO-101
* Parent(s)/legal guardian(s) of participant willing and able to complete the informed consent process and comply with study procedures and visit schedule

Exclusion Criteria:

* Planned or current participation in another clinical trial that may confound the safety and efficacy evaluation of ABO-101 during the duration of this study
* Any other situation that precludes the participant from undergoing procedures required in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This long-term follow-up study will enroll up to 24patients with MPS IIIB from prior ABO-101 clinical trials. Participants from the previous trials are of any racial, ethnic, or gender background, and could be in the early, middle or advanced phase of the disease
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 60 months
  Long-term product safety as defined by the incidence, type, and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Age Equivalent Compared to Natural History Study Data | AII study visits (30, 36, 42, 48, and 60 Months)
  Change from baseline in the Age Equivalent after treatment compared to Natural History Study data calculated by the Mullen Scales of Early Learning or the Kaufman Assessment Battery far Children; Second Edition, based on chronological and developmental age
Developmental Quotient Compared to Natural History Study Data calculated by the Mullen Scales of Early Learning or the Kaufman Assessment Battery for Children | AII study visits (30, 36, 42, 48, and 60 Months)
  Change from baseline in the Developmental Quotient (DQ) after treatment compared to Natural History Study data calculated by the Mullen Scales of Early Learning or the Kaufman Assessment Battery for Children; Second Edition, based on chronological and developmental age
Cognitive Age Equivalent Compared to Natural History Study Data | AII study visits (30, 36, 42, 48, and 60 Months)
  Change from baseline in the Cognitive Age Equivalent after treatment compared to Natural History Study, calculated using the Bayley Scales of lnfant and Toddler Development - Third edition or the Kaufman Assessment Battery far Children. Second Edition, based on developmental age
Developmental Quotient Compared to Natural History Study Data calculated using the Bayley Scales of lnfant and Toddler Development or the Kaufman Assessment Battery for Children | AII study visits (30, 36, 42, 48, and 60 Months)
  Change from baseline in the Developmental Quotient after treatment compared to Natural History Study, calculated using the Bayley Scales of lnfant and Toddler Development - Third edition or the Kaufman Assessment Battery far Children. Second Edition, based on developmental age
Adaptive Age Equivalent Compared to Natural History Study Data | AII study visits (30, 36, 42, 48, and 60 Months)
  Change from baseline in the Adaptive Age Equivalent score after treatment compared to Natural History Study data, as assessed by parent report using the Vineland Adaptive Behavior Scale II Survey farm
Pediatric Quality of Life lnventory (PedsQL ™) | AII study visits (30, 36, 42, 48, and 60 Months)
  Quality of life based on Pediatric Quality of Life lnventory (PedsQL ™) applicable for participants who completed these evaluations in the prior clinical trial.
Parenting Stress lndex, 4th Edition (PSl-4) | AII study visits (30, 36, 42, 48, and 60 Months)
  Quality of life based on Parenting Stress lndex, 4th Edition (PSl-4).
Parental Global lmpression Scale | AII study visits (30, 36, 42, 48, and 60 Months)
  Evolution on Parental Global lmpression Score, applicable for patients who completed these evaluations in the prior clinical trial.
Clinical Global lmpression lmprovement Scale | AII study visits (30, 36, 42, 48, and 60 Months)
  Evolution of Clinical Global lmpression lmprovement Score applicable for patients who completed these evaluations in the prior clinical trial.
Parent Symptom Scale Questionnaire | AII study visits (30, 36, 42, 48, and 60 Months)
  Evolution on Parent Symptom Score Questionnaire applicable for patients who completed these evaluations in the prior clinical trial.
T-cell responses against the AAV9 capsid | 60 Months
  Long-term immunological responses defined as T-cell responses against the AAV9 capsid
T-cell responses against the α-N- acetylglucosaminidase (NAGLU) transgene product | 60 Months
  Long-term immunological responses defined as T-cell responses against the α-N- acetylglucosaminidase transgene product.
Antibody formation (humoral) against the α-N- acetylglucosaminidase (NAGLU) transgene product | 60 Months
  Long-term immunological responses defined as antibody formation (humoral) against the α-N- acetylglucosaminidase (NAGLU)
Antibody formation (humoral) against the AAV9 capsid | 60 Months
  Long-term immunological responses defined as antibody formation (humoral) against the AAV9 capsid.
Viral Load | AII study visits (30, 36, 42, 48, and 60 Months)
  Long-term viral load, in applicable cases.

OTHER OUTCOMES:
Sanfilippo Behavior Rating Scale | 30, 36, 42, 48, and 60 Months
  Change from baseline in the Sanfilippo Behavior Rating Scale (SBRS) scale after treatment compared to Natural History Study data, as assessed by parent report using the Sanfilippo Behavior Rating Scale form. Minimum value is 0 and maximum value is 6 where higher score indicates a worse outcome
Children's Sleep Habits Questionnaire (CSHQ) | 30, 36, 42, 48, and 60 Months
  Quality of life based on sleep-pattern evaluation based on modified Children's Sleep Habits Questionnaire (CSHQ).Minimum value is 1 and maximum value is 111 where higher scores indicates a worse outcome
Neutralizing antibody against the AAV9 capsid | 60 Months
  Long-term immunological responses defined as neutralizing antibody formation against the AAV9 capsid

CONTACTS AND LOCATIONS:
Locations (3):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- Armand-Trousseau Hospital, Paris, France
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data